CLINICAL TRIAL: NCT03280277
Title: Novel Imaging of Lymph Nodes in Patients With Rectal Cancer Using Ferumoxytol Enhanced MRI
Brief Title: Ferumoxytol-Enhanced MRI in Imaging Lymph Nodes in Patients With Locally Advanced Rectal Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); Radiological Society of North America (Other)
Responsible Party: Principal Investigator, Alexander Guimaraes, Associate Professor, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00016101; NCI-2017-00388 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ONC-16108-L; STUDY00016101 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2017-05-23; First posted 2017-09-12 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Locally Advanced Rectal Carcinoma; Stage III Rectal Cancer AJCC v7; Stage IIIA Rectal Cancer AJCC v7; Stage IIIB Rectal Cancer AJCC v7; Stage IIIC Rectal Cancer AJCC v7
MeSH Terms: conditions — Rectal Neoplasms | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (ferumoxytol-enhanced MRI) (Experimental): Patients receive ferumoxytol IV over 15 minutes and then after 24-36 hours undergo ferumoxytol-enhanced MRI before start of neoadjuvant therapy and within 4 weeks before surgery.
  Interventions: Procedure: Contrast-enhanced Magnetic Resonance Imaging; Drug: Ferumoxytol

INTERVENTIONS:
Procedure: Contrast-enhanced Magnetic Resonance Imaging — Undergo ferumoxytol-enhanced MRI
  Other Names: CONTRAST ENHANCED MRI; Contrast-enhanced MRI
Drug: Ferumoxytol — Given IV
  Other Names: Feraheme; Ferumoxytol Non-Stoichiometric Magnetite

SUMMARY:
This pilot clinical trial studies how well ferumoxytol-enhanced magnetic resonance imaging (MRI) works in imaging lymph nodes in patients with rectal cancer that has spread from where it started to nearby tissue or lymph nodes (locally advanced). Ferumoxytol is a form of very small iron particles that are taken up by cells in normal lymph nodes and may work better in imaging patients with rectal cancer when given with MRI.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine feasibility of administering ferumoxytol and obtaining ferumoxytol enhanced magnetic resonance (MR) images in patients with resectable locally advanced rectal cancer with enlarged or suspicious lateral pelvic lymph nodes before starting neoadjuvant therapy and again before total mesorectal excision.

SECONDARY OBJECTIVES:

I. To collect detailed information about the location of ultrasmall superparamagnetic iron oxide (USPIO)-MRI detected lymph nodes prior to neoadjuvant therapy and again prior to total mesorectal excision.

II. To compare the sensitivity and specificity of ferumoxytol enhanced MR imaging in assessment of pathological lymph nodes with those of non-USPIO-MRI and positron emission tomography-computed tomography (PET-CT).

OUTLINE:

Patients receive ferumoxytol intravenously (IV) over 15 minutes and then after 24-36 hours undergo ferumoxytol-enhanced MRI before start of neoadjuvant therapy and within 4 weeks before surgery.

After completion of study treatment, patients are followed up for 4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed, locally advanced, malignancy of the rectum; based on multi-disciplinary tumor board discussion, patients are candidates for tri-modality treatment
* Stage T1-4bN1-2, by the American Joint Committee on Cancer (AJCC) 7th edition, based on the following minimum workup:

  * CT chest/abdomen with contrast
  * MRI pelvis with contrast
  * PET/CT of the whole-body or skull base to mid-thigh
* Subjects must have had no prior therapy for cancer of the rectum
* Members of all races and ethnic groups will be included
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* White blood cell count >= 3.0 K/cu mm
* Absolute neutrophil count >= 1.5 K/cu mm
* Platelets >= 100 K/cu mm
* Hemoglobin >= 8.0 g/dl (the use of transfusion or other invention to achieve hemoglobin [Hgb] >= 8.0 g/dl is acceptable)
* Total bilirubin =< 1.5 X institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for subjects with creatinine levels above institutional normal
* Woman of childbearing potential, a negative serum or urine pregnancy test
* Willingness to use adequate contraception for 12 months after completion of all therapy
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Subjects with AJCC 7th edition stage TxN0 and/or metastatic disease outside of pelvis (suspicious lateral pelvic lymph nodes up to and including common iliacs are allowed on the protocol)
* Prior systemic chemotherapy for rectal cancer; prior chemotherapy for another malignancy is allowable as long as it has been > 2 years since completion of therapy for previous malignancy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ferumoxytol or other agents used in the study
* Prior abdominopelvic radiation or radiation for rectal cancer
* History of other malignancy in the past 2 years except non-melanomatous skin cancer, breast ductal carcinoma in situ (DCIS) and low-risk prostate adenocarcinoma
* Medical contraindications to low anterior resection or abdominoperineal resection
* Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because chemoradiotherapy has the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to the use of ferumoxytol as a contrast agent in the mother, breastfeeding should be discontinued if the mother receives ferumoxytol while nursing; men who are sexually active and not willing/able to use medically acceptable forms of contraception are also excluded from this study
* Subjects with multiple drug allergies and/or subjects who have had an allergic reaction to any intravenous iron replacement product or a known history of hypersensitivity to ferumoxytol
* Subjects with concurrent clinical diagnosis of evidence of active iron overload defined by the following 1) ferritin >= 250 ng/mL in men or >= 200 ng/mL in women AND 2) transferrin saturation, the ratio of plasma iron to transferrin, expressed as percent, >= 45%
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ferumoxytol
* Patients with renal insufficiency; glomerular filtration rate (GFR) < 60
* Adult patients who require monitored anesthesia for MRI scanning
* Subjects who have a contraindication for MRI: metal in their bodies (a cardiac pacemaker or other incompatible device), are severely agitated, or have an allergy to gadolinium (Gd) contrast material
* Subjects with known hepatic insufficiency or cirrhosis as determined by either a prior diagnosing physician or at review at initial consultation; these disease entities do not have formal associated lab values and are thus a clinical diagnosis by the prior aforementioned physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
Practical feasibility | Up to 6 weeks
  Assessed by successful accrual objectively, as a percentage of all subjects enrolled. Accrual success will be measured in binary fashion; successful accrual is considered a patient that enrolls and completes the entire trial. All other eligible patients will be considered an accrual failure. Practical feasibility will be considered a success if greater than 50%.
Technical feasibility of ultrasmall superparamagnetic iron oxide (USPIO) - magnetic resonance imaging (MRI) of the chest | Up to 6 weeks
  Assessed by image quality and protocol completion. Will be evaluated in a descriptive manner. Image quality, readability (i.e. the ability for diagnostic radiologist to make an appropriate diagnostic conclusion), completion of ferumoxytol infusion, data acquisition, and completion of magnetic resonance protocol.

SECONDARY OUTCOMES:
Reason for accrual failure | Up to 6 weeks
Report location and enhancement patterns on USPIO - MRI | Up to 6 weeks
Sensitivity and specificity of MRI imaging for all lymph nodes | Up to 6 weeks
  Assessed by pathology finding. Sensitivities and specificities of ferumoxytol enhanced MRI prior to neoadjuvant therapy will be calculated using pathology finding as the gold standard. Each lymph node will be treated as an independent observation. The sensitivity and specificity will be compared with those from positron emission tomography (PET)/computed tomography (CT) findings using McNemar's test. Sensitivities and specificities of ferumoxytol enhanced MRI before surgery will also be calculated as a reference.
Sensitivity and specificity of PET/CT imaging | Up to 6 weeks
  Assessed by pathology finding. Sensitivities and specificities of ferumoxytol enhanced MRI prior to neoadjuvant therapy will be calculated using pathology finding as the gold standard. Each lymph node will be treated as an independent observation. The sensitivity and specificity will be compared with those from PET/CT findings using McNemar's test. Sensitivities and specificities of ferumoxytol enhanced MRI before surgery will also be calculated as a reference.
Accuracy of USPIO - MRI | Up to 6 weeks
  Accuracy, which is defined as the percentage of all patients or lymph nodes in which MRI with ferumoxytol correctly predicted the presence or absence of metastatic tumor, will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Guimaraes, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States